CLINICAL TRIAL: NCT00735683
Title: Double-Blind, Randomized, Placebo-Controlled, 12-Week Study of the Safety and Efficacy of ATHX-105 Phosphate for the Treatment of Obesity
Brief Title: A Short-Term Study to Examine the Effects of ATHX-105 Phosphate on Weight Loss and Safety
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Dr. John J. Harrington, Chief Scientific Officer, Athersys Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01-03
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: Weight loss; Weight-loss drugs; Obesity; Overweight; Body weight; Diet; Metabolic Disorder; Nutrition Disorder
MeSH Terms: conditions — Obesity; Weight Loss; Overweight; Body Weight; Metabolic Diseases; Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: ATHX-105 phosphate
- 3 (Experimental)
  Interventions: Drug: ATHX-105 phosphate
- 4 (Experimental)
  Interventions: Drug: ATHX-105 phosphate
- 5 (Experimental)
  Interventions: Drug: ATHX-105 phosphate
- 6 (Experimental)
  Interventions: Drug: ATHX-105 phosphate

INTERVENTIONS:
Drug: ATHX-105 phosphate — includes diet, physical activity, and lifestyle modification
  Arms: 2; 3; 4; 5; 6
Drug: Placebo — includes diet, physical activity, and lifestyle modification
  Arms: 1

SUMMARY:
This primary purpose of this study is to determine if ATHX-105 phosphate causes weight loss over a 12-week period.

DETAILED DESCRIPTION:
The rate of obesity in adults continues to increase. Obesity affects overall health and is associated with an increased risk for diabetes, high blood pressure, coronary artery disease, osteoarthritis, and sleep apnea. To date, the medication options to treat obesity have been limited.

This study will examine if a new investigational drug, ATHX-105 phosphate, may cause weight loss in humans over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults with a body mass index of 30-45 kg/m2

Exclusion Criteria:

* Pregnancy
* Diabetes
* Adults with serious or unstable current or past medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | 12 weeks

SECONDARY OUTCOMES:
vital signs, lipids/glucose, waist circumference | 12 weeks